CLINICAL TRIAL: NCT02378363
Title: Representations and Prevention of Cancers in Schools
Acronym: RISCOLAIRE
Status: Completed | Type: Observational
Sponsor: Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-03
Record Dates: First submitted 2015-02-06; First posted 2015-03-04 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-02

CONDITIONS: Healthy
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Student 9 to 12 years: Students aged 9 to 12 years and enrolled in classes CM1, CM2 and 6th
  Interventions: Other: Write, draw and interview

INTERVENTIONS:
Other: Write, draw and interview — Child should write, draw cancer signifiance and after, they were interview by a school nurse about cancer signifiance.

SUMMARY:
The main objective is to develop an educational program and to measure the impact on social representations identified as acting in the prevention of cancer. Child should write, draw and speak about cancer signifiance to identify individual conceptions and representations of health and cancer in children aged 9 to 12 years in school.

DETAILED DESCRIPTION:
The stages are :

* Selection of forms
* Technique of write and draw and interview by a school nurse
* Data analysis

ELIGIBILITY:
Inclusion Criteria:

* Aged between 9 and 12

Exclusion Criteria:

* Boy or Girl ages over 12 years and under 9 years
* Children refusal

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: students aged 9 to 12 years and enrolled in classes CM1, CM2 and 6th
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2012-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Number of cancer and health representations in children | 60 minutes
  Identification of individual cancer and health conceptions and representations in children aged 9 to 12 years in schools

SECONDARY OUTCOMES:
Number of association of cancer and health representations with the ecological deprivation index | 60 minutes
  Assess whether the prevalence of cancer and health representations is associated with socioeconomic level school zones

CONTACTS AND LOCATIONS:
Overall Officials: Franck Chauvin, PhDMD, Study Director — ICLN